CLINICAL TRIAL: NCT02342223
Title: Voluma Treatment of HIV Facial Lipoatrophy
Brief Title: Voluma Filler Agent For The Treatment of HIV-associated Facial Lipoatrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jared Jagdeo, MD, MS (U.S. Federal Agency)
Collaborators: Allergan (Industry); VA Northern California Health Care System (U.S. Federal Agency); East Bay Institute for Research and Education (Other)
Responsible Party: Sponsor-Investigator, Jared Jagdeo, MD, MS, Medical Physician, VA Northern California Health Care System
Organization: VA Northern California Health Care System (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allergan-97727
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: HIV Facial Lipoatrophy
Keywords: human immunodeficiency virus; facial lipoatrophy; facial lipodystrophy; hyaluronic acid; dermal filler; filler agent
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voluma (Experimental): Subjects will be screened for severity on their HIV facial lipoatrophy according to the Carruthers Lipoatrophy Severity Scale (CLSS), and will receive subcutaneous injections of Voluma in the affected facial areas with the 'smile and fill' technique (Jagdeo 2014) based on Carruthers scoring scale.
  Subjects with Carruthers Score level 2 will receive total of 2-6 syringes of Voluma.
  Subjects with Carruthers Score level 3 will receive total of 4-8 syringes of Voluma.
  Subjects with Carruthers Score level 4 will receive total of 6-12 syringes of Voluma.
  All subjects will receive one Voluma treatment at initial time = 0 and may be eligible for touchup treatment, if necessary, at 2 weeks post-initial treatment.
  Interventions: Device: Voluma

INTERVENTIONS:
Device: Voluma
  Other Names: 20 mg/ml hyaluronic acid-based dermal filler

SUMMARY:
The purpose of this study is to test the safety of Voluma and see what effects it has on HIV facial lipoatrophy. The hypothesis is that Voluma will be safe, efficacious and positively impact the quality-of-life in the treatment of facial lipoatrophy in patients with HIV.

DETAILED DESCRIPTION:
HIV facial lipoatrophy (volume loss) is an increasing concern with patients on Highly Active Anti-Retroviral Therapy (HAART) because it affects the quality-of-life and adherence to medication regimen. Treatment of HIV facial lipoatrophy helps to improve patient wellness by removing the social stigma associated with HIV facial lipoatrophy. Currently, there are few medical therapies that can treat HIV facial lipoatrophy and are FDA-approved for this indication. Juvéderm Voluma (Allergan) may benefit patients on HAART because it may provide a more immediate aesthetic enhancement and potentially has fewer adverse effects, which results in a more natural appearing facial enhancement outcome. Voluma is the only agent that is FDA-approved for facial volume loss. We anticipate Voluma having less adverse effects than current FDA-approved drugs for HIV lipoatrophy as Voluma is a hyaluronic acid (HA)-based agent. The benefit of using hyaluronidase to "correct" or "modify" facial HA-based volume therapy is also a benefit for HIV patients, which currently does not exist as a post-injection modification option for other FDA-approved filling agents used to treat patients with HIV facial lipoatrophy. Voluma is currently FDA-approved for correction of age-related volume loss in the midface, and there's no alteration in the chemical or biophysical properties of Voluma that is being used in our proposed study. In addition to conventional injection techniques, we will implement the 'smile and fill' technique pioneered by our clinical research group to achieve better mid-face aesthetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more with laboratory evidence of HIV-1 infection and have been on HAART therapy for at least 1 (one) year.
* Not to have AIDS (CD4 count < 250) or AIDS-defining illness.
* Bilateral lipoatrophy corresponding to a visual grade 2 or above in the attached Carruthers Lipoatrophy Severity Scale (CLSS).
* Available and willing to attend study follow-up visits.
* Able and willing to give informed consent.

Exclusion Criteria:

* Any active skin inflammation or infection in or near the treatment area.
* Hypersensitivity to the components of Voluma.
* Previous treatment with Voluma or any other product for facial lipoatrophy within the past year.
* Has known bleeding disorder
* History of keloid formation
* Currently receiving systemic corticosteroids or anabolic steroids
* Currently on known anticoagulants (i.e. aspirin, non-steroidal anti-inflammatory drugs)
* Pregnancy or breastfeeding or anticipating becoming pregnant during the study period.
* Any other excluding factors that, according to the investigator's judgment, would preclude enrollment in the study.
* Any condition that may interfere with ability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Jagdeo, MD, MS, Principal Investigator — Sacramento VA Medical Center - Dermatology Service
Locations (1):
- Sacramento VA Medical Center, Mather, California, United States

REFERENCES:
- [Result] Wang AS, Babalola O, Jagdeo J. The "smile-and-fill" injection technique: a dynamic approach to midface volumization. J Drugs Dermatol. 2014 Mar;13(3):288-90. PMID 24595573
- [Result] Bechara FG, Gambichler T, Brockmeyer NH, Sand M, Altmeyer P, Hoffmann K. Hyaluronic acid new formulation: experience in HIV-associated facial lipoatrophy. Dermatology. 2008;217(3):244-9. doi: 10.1159/000148252. Epub 2008 Jul 25. PMID 18663308
- [Derived] Ho D, Jagdeo J. Patient Reported Outcomes from HIV Facial Lipoatrophy Treatment With a Volumizing Hyaluronic Acid Filler: A Prospective, Open-Label, Phase I and II Study. J Drugs Dermatol. 2016 Sep 1;15(9):1064-9. PMID 27602967

RESULTS

PARTICIPANT FLOW:
Groups:
- Voluma Treatment of HIV Facial Lipoatrophy: Subjects were screened for severity on their HIV facial lipoatrophy according to the Carruthers Lipoatrophy Severity Scale (CLSS), and received subcutaneous injections of Voluma in the affected facial areas with the "smile and fill" technique (Jagdeo 2014) based on Carruthers scoring scale.
  All subjects received one Voluma treatment at initial time = 0 and may be eligible for touchup treatment, if necessary, at 2 weeks post-initial treatment.
Period: Overall Study
Arm/Group | Voluma Treatment of HIV Facial Lipoatrophy
Started | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Voluma: Subjects were screened for severity on their HIV facial lipoatrophy according to the Carruthers Lipoatrophy Severity Scale (CLSS), and received subcutaneous injections of Voluma in the affected facial areas with the "smile and fill" technique (Jagdeo 2014) based on Carruthers scoring scale.
  All subjects received one Voluma treatment at initial time = 0 and may be eligible for touchup treatment, if necessary, at 2 weeks post-initial treatment.
Arm/Group | Voluma
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Rated Very Much Improved on the Global Aesthetic Improvement Scale (GAIS) by Prinicple Investigator
Description: To evaluate the effectiveness of Voluma injections as a treatment for HIV-associated facial lipoatrophy over 12 months by assessing changes in the Global Aesthetic Improvement Scale (GAIS) based on pre- and post-treatment photography by principal investigator (PI). GAIS is a 5-point rating scale, ranging from "worse, no change, improved, much improved, and very much improved."
Time Frame: Baseline to 12 months
Measure: Number; unit: participants
Arm/Group | Voluma
Number analyzed (Participants) | 19
participants | 19

2. Primary Outcome: Percentage of Participants With Device or Procedure Related Adverse Events
Description: To evaluate the safety of Voluma injections as a treatment for HIV-associated facial lipoatrophy over 12 months by monitoring the incidence of adverse events (patient will keep a daily diary for initial 1 month and weekly phone calls will be made by study coordinator for initial 1 month to document possible adverse events, including injection site reactions, redness, bruising, swelling, and induration).
Time Frame: 12 months
Population: Common, transient adverse events reported in subject diaries include as follows.
Measure: Number; unit: percentage of total participants
Arm/Group | Voluma
Number analyzed (Participants) | 19
percentage of total participants
  Ecchymosis | 42
  Edema | 47
  Tenderness | 21
  Pain | 42
  Permanent Treatment Related AE | 0

3. Secondary Outcome: Number of Participants Achieving Grade 1 in the Carruthers Lipoatrophy Severity Scale (CLSS)
Description: To evaluate the effectiveness of Voluma injections as a treatment for HIV-associated lipoatrophy over 12 months by assessing changes in the Carruthers Lipoatrophy Severity Scale (CLSS) based on pre/post intervention photography by principal investigator (PI). CLSS is a 4-point grading scale (1 to 4, with a greater number indicating higher severity of HIV FLA). Grade 1: mild and localized facial lipoatrophy. Grade 2: deeper and longer atrophy, with the facial muscles beginning to show through. Grade 3: atrophic area is even deeper and wider, with the muscles clearly showing. Grade 4: lipoatrophy covers a wide area, extending up toward the eye sockets, and the facial skin lies directly on the muscles.
Time Frame: Baseline to 12 months
Measure: Number; unit: Participants
Arm/Group | Voluma
Number analyzed (Participants) | 19
Participants | 19

4. Secondary Outcome: Number of Participants Rated Very Much Improved on the Global Aesthetic Improvement Scale (GAIS) by Participants
Description: To evaluate the effectiveness of Voluma injections as a treatment for HIV-associated facial lipoatrophy over 12 months by assessing changes in the Global Aesthetic Improvement Scale (GAIS) based on pre- and post- treatment photography by participants.
Time Frame: Baseline to 12 months
Measure: Number; unit: Participants
Arm/Group | Voluma
Number analyzed (Participants) | 19
Participants | 19

5. Secondary Outcome: Subject Satisfaction Questionnaire (SSQ)
Description: To evaluate the benefits and effects of Voluma injections on HIV-associated facial lipoatrophy as evidenced by the subject satisfaction questionnaire.
Time Frame: 12 months
Measure: Number; unit: percentage of total participants
Arm/Group | Voluma
Number analyzed (Participants) | 19
percentage of total participants
  "Has this treatment been beneficial to you?" | 100
  "Would you get this treatment again?" | 100
  "Would you recommend this treatment to others?" | 100

6. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: To evaluate the effects of Voluma injections on the subject's quality of life (QOL) using the Dermatology Life Quality Index (DLQI). The DLQI is a validated 10-item questionnaire encompassing six different domains of QOL, including symptoms and feelings, daily activities, leisure, work/school, personal relationships, and treatment. Each question has four possible responses: "not at all/not relevant," "a little," "a lot," and "very much" that corresponds to scores of 0, 1, 2, and 3, respectively, and a higher score suggests a higher level of QOL impairment. DLQI total score may range between 0 to 30.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Voluma
Number analyzed (Participants) | 19
scores on a scale
  Baseline | 1.6 (3.0)
  12-months post-treatment | 0.5 (1.2)

ADVERSE EVENTS:
Description: Common, transient adverse events were documented and reported in subject diaries.
Arm/Group | Voluma
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 9/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voluma (N=19)
Ecchymosis (Injury, poisoning and procedural complications) | 8 (19)
Edema (Injury, poisoning and procedural complications) | 9 (19)
Tenderness (Injury, poisoning and procedural complications) | 4 (19)
Pain (Injury, poisoning and procedural complications) | 8 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No